CLINICAL TRIAL: NCT03376750
Title: Effectiveness of a Tele-rehabilitation Intervention to Improve Performance and Reduce Morbidity for People Post Hip Fracture - Randomized Controlled Trial
Brief Title: Tele-rehabilitation Intervention for People Post Hip Fracture - Randomized Controlled Trial (RCT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Herzog Hospital (Other)
Collaborators: Hebrew University of Jerusalem (Other); Israel National Institute for Health Policy and Health Services Research (Other Government)
Responsible Party: Principal Investigator, Yakir Kaufman, MD, Herzog Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HerzogH RCT
Record Dates: First submitted 2017-12-13; First posted 2017-12-18 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Hip Fractures
Keywords: telerehabilitation; occupational therapy; RCT; participation; quality of life; intervention; older adults
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: three-arm randomized control trail (RCT) including pre/post intervention and follow-up
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CO - OP via telerehabilitation + standard care (Experimental): 10 CO-OP videoconferencing sessions from an occupational therapist . Each session will be utilized to guide the participants to achieve their self-identified goals, focusing on problem-solving for daily life situations and on the ability to implement the discussed strategies for a variety of activities.
  Interventions: Behavioral: CO - OP
- CO - OP via face to face + standard care (Experimental): 10 CO - OP face to face sessions from an occupational therapist. Each session will be utilized to guide the participants to achieve their self-identified goals, focusing on problem-solving for daily life situations and on the ability to implement the discussed strategies for a variety of activities.
  Interventions: Behavioral: CO - OP
- control group - standard care (No Intervention): standard care as given from public health service

INTERVENTIONS:
Behavioral: CO - OP — CO-OP is a top-down, task-oriented, client-centered approach that uses an iterative process of dynamic performance analysis and guided discovery to enable individuals to identify strategies that will improve performance
  Other Names: Cognitive Orientation to Occupational Performance
  Arms: CO - OP via face to face + standard care; CO - OP via telerehabilitation + standard care

SUMMARY:
Most surviving hip-fracture patients experience reduced mobility and lose their functional ability, which increases the risk of complications and rehospitalization. Post-discharge transitional programs to reduce readmissions have shown some success. Telerehabilitation refers to the use of technologies to provide rehabilitation services to people in their homes. Considering the need for long-term follow-up care for people with hip fracture, in-home telerehabilitation could increase independence, decrease hospital stays and reduce the burden for caregivers.

The purpose of this three armed randomized controlled trial is to investigate the effectiveness of an intervention program based on telerehabilitation on ADL, QOL, depression and burden on caregivers compared to face-to-face home visits and usual care of community-dwelling older adults after hip fracture.

90 older people with hip fractures will be randomly assigned to a telerehabilitation group (N=30), face-to-face visits (N=30) and a control group.

The aim of the intervention is to improve the transition from rehabilitation units to community dwelling. It will include 10 videoconferencing/ face-to-face sessions from an occupational therapist in the presence of the primary caregiver. Each session will be utilized to guide the participants to achieve their self-identified goals, focusing on problem-solving for daily life situations and on the ability to implement the discussed strategies for a variety of activities

ELIGIBILITY:
Inclusion Criteria:

Older adults (age ≥60 years) post hip fracture - discharged from the inpatient rehabilitation unit of Herzog Hospital, Jerusalem, between January 2017 and December 2017.

Discharge from rehabilitation to a non-institutionalized setting. broadband or Wi-Fi in their home and must be able to operate an iPad independently.

FIM>90 at discharge. Has a designated caregiver (a close friend, family member, or support worker) aged over 18, and a Hebrew, English or Arabic speaker, who will agree to cooperate in the research

Exclusion Criteria:

Aphasia. cognitive impairment (Montreal Cognitive Assessment scores : MOCA<19 or MMSE<21).

degenerative neurological diagnoses. current major depressive or psychotic disorder. other acute or chronic health condition that will influence their ability to participate in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline at post intervention in The Canadian Occupational Performance Measure (COPM) | Baseline-pretest (T0), immediately following intervention (post intervention 10 weeks) (T1), and a 6-month follow-up (T2). in total, 9 months
  The COPM will be used for measuring performance and satisfaction with personally identified participation goals. Participants are asked to identify goals and then rate their performance and satisfaction with current status on a scale from 1 to 10, where 10 indicates optimal performance or satisfaction

SECONDARY OUTCOMES:
Functional Independence Measure (FIM) | Baseline-pretest (T0), immediately following intervention (post intervention 10 weeks) (T1), and a 6-month follow-up (T2). in total, 9 months
  The aim of the FIM is to monitor the recovery of functional ability by people undergoing rehabilitation. The FIM is comprised of 18 parameters, each rated on a scale of 1-7 (range = 18-126) according to the degree of assistance required to perform a specific activity
The Geriatric Depression Scale (GDS) | Baseline-pretest (T0), immediately following intervention (post intervention 10 weeks) (T1), and a 6-month follow-up (T2). in total, 9 months
  The scale consists of 15 items; each item has two possible answers (yes or no). The highest possible score is 15, which indicates the most severe depressive state.
12-item MOS Short-Form Health Status Survey, Hebrew version | Baseline-pretest (T0), immediately following intervention (post intervention 10 weeks) (T1), and a 6-month follow-up (T2). in total, 9 months
  This generic HR-QoL instrument focuses on functional status. The questionnaire includes 12 items taken directly from the SF-36[73] which are used to calculate the Physical and Mental Component Summary. The first question measured by the SF-12 is an acceptable self-rated measure for general health
The Zarit Caregiver Burden Interview | Baseline-pretest (T0), immediately following intervention (post intervention 10 weeks) (T1), and a 6-month follow-up (T2). in total, 9 months
  The ZBI includes 22 statements recorded in a 0-4 Likert scale (total score range 0 to 88, where higher scores mean higher burden), which rates the subjective component of burden
Qualitative interview | post intervention, 10 weeks (T1)
  Semi-structured interviews will be conducted post intervention with the patients and their caregivers to identify barriers and facilitators regarding the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Yafit Gilboa, OTphD, Study Director — School of Occupational Therapy, Faculty of Medicine Hadassah and the Hebrew University of Jerusalem
Locations (1):
- Herzog Hospital, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gilboa Y, Maeir T, Karni S, Eisenberg ME, Liebergall M, Schwartz I, Kaufman Y. Effectiveness of a tele-rehabilitation intervention to improve performance and reduce morbidity for people post hip fracture - study protocol for a randomized controlled trial. BMC Geriatr. 2019 May 20;19(1):135. doi: 10.1186/s12877-019-1141-z. PMID 31109289